CLINICAL TRIAL: NCT01453920
Title: Choroidal Neovascular Membrane Recurrence Rate in Wet AMD Patients Stable on Three Month Ranibizumab Dosing
Brief Title: Wet AMD Recurrence Rate in Patients Stable on Three Month Ranibizumab Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0686-AE
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Age Related Macular Degeneration
Keywords: Age Related Macular Degeneration; Choroidal Neovascular Membrane
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treat-and-extend (Active Comparator): Ranibizumab injection every 3 months, with follow-up assessments at each visit (every 3 months)
  Interventions: Drug: Ranibizumab
- Treat-and-observe' (Experimental): No injection, follow-up assessments every month
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal Ranibizumab 0.05cc (10mg/ml)
  Other Names: Lucentis
  Arms: Treat-and-extend
Drug: Ranibizumab — Intravitreal Ranibizumab 0.05cc (10mg/ml)
  Other Names: Lucentis
  Arms: Treat-and-observe'

SUMMARY:
The current norm in clinical practice for the treatment of choroidal neovascular membranes (CNVM) secondary to Age-related Macular Degeneration(AMD) involves monthly injections of Ranibizumab until the disease is stabilized. At this point, most physicians tend to follow one of two treatment regimens. 'Treat -and-observe' entails regular follow-up of stable patients, with treatment thereafter only in the presence of disease recurrence. Alternatively, in a 'treat-and-extend' dosing strategy, intervals between treatments are extended as long as disease remains stable. Many clinicians, who employ a treat-and-extend dosing regimen, do not extend their treatment intervals beyond 3 months. However, it is possible that the subgroup of patients on every three months 'treat-and-extend' dosing may represent a uniquely, stable population that would perform particularly well on an observational regimen with regular follow-up. We hypothesize that there will be a low CNVM recurrence rate in wet AMD patients stable on every three months Ranibizumab dosing ('treat-and-extend'), who begin a treat-and-observe protocol.

DETAILED DESCRIPTION:
In North America, AMD is the leading cause of irreversible vision loss in those over 65 years of age.1 Vascular endothelial growth factor A (VEGF-A) is a potent promoter of angiogenesis and vascular permeability and its role in the pathogenesis of neovascular AMD is well recognized.2,3 The advent of VEGF inhibitors such Ranibizumab (Lucentis; Genentech Inc.) has revolutionized the management of neovascular AMD. Ranibizumab is an intravitreally administered recombinant, humanized, monoclonal antibody antigen-binding fragment (Fab) that neutralizes all known active forms of VEGF-A. In the landmark phase III clinical studies MARINA, and ANCHOR, Ranibizumab injections were administered monthly over the course of 2 years to eyes with subfoveal CNVMs secondary to AMD. Ranibizumab was shown to not only prevent loss of visual acuity (VA) but also improve VA on average in these patients. 4-6

Despite the tremendous benefit of this treatment, the prospect of indefinitely adhering to the monthly treatment schedules of MARINA and ANCHOR has raised ocular and systemic safety concerns as well as convenience and cost issues for patient and physician alike. The identification of alternative dosing strategies capable of reducing the number of required anti-VEGF injections while still achieving favourable visual acuity outcomes has since been a subject of great interest. The current norm in clinical practice with Ranibizumab is to implement an 'initiation phase' followed by an individualized 'maintenance phase' that is modeled after one of two basic approaches: 'treat-and-observe' or 'treat-and-extend'. Both regimens are currently considered within the standard of clinical practice. 'Treat -and-observe' entails treatment and follow-up until the macula is free of exudation, with treatment thereafter only in the presence of recurrent exudation.7 Alternatively, in a treat-and-extend dosing strategy, intervals between treatments are extended as long as the macula remains dry.8 In the 2009 ASRS survey, 56% of physicians reported employing treat-and-observe and 44% reported employing treat-and-extend for their patients with neovascular AMD.9 In a study by Oubraham et al10 it was found that a treat-and-extend dosing regimen may yield greater gains in vision than treat-and-observe, albeit with a greater number of required injections.

In a treat-and-extend dosing strategy, some patients may require frequent monthly injections to stabilize their disease, while others may demonstrate a more stable condition requiring infrequent treatments. Many clinicians who employ a treat-and-extend dosing regimen, do not extend their treatment intervals beyond 3 months. However, it is possible that the subgroup of patients on every three months 'treat-and-extend' dosing may represent a unique, stable population that would perform particularly well on a 'treat-and-observe' regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or more
* Active primary or recurrent choroidal neovascularization secondary to AMD in the study eye, currently stable on an 'every three month' treatment regimen (established using a treat and extend dosing protocol)
* Best-corrected visual acuity of Counting Fingers or better (Snellen equivalent) in the study eye
* All IVFA lesion types and lesion sizes
* One eye per subject (the "study eye"). If both eyes are eligible, the one with better VA will be selected unless, for medical reasons, the other is more appropriate

Exclusion Criteria:

* Treatment of the current choroidal neovascular membrane with verteporfin photodynamic therapy (PDT), external-beam radiation therapy, transpupillary thermotherapy, or subfoveal laser photocoagulation (or juxtafoveal or extrafoveal laser photocoagulation
* History of vitrectomy surgery in the study eye
* Individuals with choroidal neovascularization from causes other than AMD

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of CNVM recurrence | 6 months
  To determine the prevalence of CNVM recurrence in each study group as defined by visual acuity (VA), dilated fundus exmaination (DFEx), Spectral Domain Optical Coherence Tomography (SDOCT) +/- Intravenous Flourescein Angiography (IVFA).

SECONDARY OUTCOMES:
Mean change in VA between baseline | 6 months
Proportion of patients losing > 15 letters (3 lines) from baseline | 6 months
Number of Ranibizumab injections | 6 months
Presence of subretinal and/or intraretinal fluid on SDOCT | 6 months
Central Retinal Thickness measurement on SDOCT | 6 months
Incidence of ocular and systemic adverse events | 6 months
Patient's sensitivity in subjectively detecting CNVM recurrence (gold standard for comparison, clinical presentation including DFEx, OCT, +/- IVFA) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Brent, MD FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada